CLINICAL TRIAL: NCT07175311
Title: Vascular Changes Associated With Endophthalmitis.
Status: Recruiting | Type: Observational
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Other Study IDs: RE-24-26
Record Dates: First submitted 2025-07-29; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Endophthalmitis
Keywords: Postoperative endophthalmitis; Multimodal imaging
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multimodal imaging findings — Fundus photography, Optical Coherence Tomography, and Fluorescein Angiography will be performed 7 days after meeting the criteria for inactivation of endophthalmitis, as outlined in the MEX-ESG guidelines. These imaging tests will be repeated one month after meeting the inactivation criteria.

SUMMARY:
This study aims to describe and investigate vascular changes associated with exogenous endophthalmitis, as well as to create a photo library where they are evidenced

DETAILED DESCRIPTION:
The implementation of multimodal imaging studies during the diagnosis and follow-up of patients with endophthalmitis may help identify, characterize, and differentiate between changes associated with host immune response, drug toxicity, or ischemia, thereby opening the possibility of implementing early treatments that lead to a better final prognosis. It is designed as a Prospective, Longitudinal, Observational, and Descriptive study. The population will be patients of the retina and vitreous service of Asociación para Evitar la Ceguera en México, who have a complete clinical record (age, sex, pathological personal history, non-pathological personal history, heredofamilial history, ophthalmologic history, allergies, medications, ophthalmologic examination with visual acuity, intraocular pressure at each visit), signed informed consent and with a history of exogenous or endogenous endophthalmitis with clear resolution criteria and clear means one week and one month after meeting the resolution criteria to be able to perform fluorescein angiography at both visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of endophthalmitis Diagnosis of Endophthalmitis
* Clinical symptoms: Pain, decrease in visual acuity, anterior chamber cells and/or vitreous turbidity, corneal edema, conjunctival hyperemia
* Laboratory studies: B-mode USG and or positive culture
* Patients who meet the endophthalmitis resolution criteria of the Mexican Endophthalmitis Study Group
* Patients with previously signed informed consent

Exclusion Criteria:

* Patients who have not signed the informed consent
* Patients under 18 years.
* Patients with endophthalmitis who do not meet the resolution criteria of the Mexican Endophthalmitis Study Group

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will be patients of the retina and vitreous service of Asociación para Evitar la Ceguera en México, who have a complete clinical record (age, sex, pathological personal history, non-pathological personal history, heredofamilial history, ophthalmologic history, allergies, medications, ophthalmologic examination with visual acuity, intraocular pressure at each visit), signed informed consent and with a history of exogenous or endogenous endophthalmitis with clear resolution criteria and clear means one week and one month after meeting the resolution criteria to be able to perform fluorescein angiography at both visits.
Sampling Method: Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Best-Corrected Visual Acuity (BCVA) | The assessment will be performed at each visit (7 days and 1 month after meeting the inactivation criteria for endophthalmitis).
  Best-Corrected Visual Acuity (BCVA) will be assessed according to the ETDRS guidelines. The test must be performed with the patient positioned 4 meters from the backlit panel, which must be calibrated to emit 85 cd/m². This procedure will be carried out by the retina fellow assigned to the case.

SECONDARY OUTCOMES:
Fluorescein Angiography | The procedure may be performed at all study visits (7 days and 1 month after meeting the inactivation criteria for endophthalmitis).
  Fluorescein angiography will be performed subsequently to evaluate associated vascular changes. The patient must undergo an 8-hour fast and have pupillary dilation with TP Ofteno® (tropicamide 5% / phenylephrine 0.8%). The procedure involves preparing the patient with aseptic technique for an intravenous injection of fluorescein dye in an upper limb, followed by imaging with a fundus camera. It is not essential to use a device of a specific brand or model, as long as a system with equivalent specifications is used consistently for the same patient throughout the study. A technician or delegated personnel may perform the procedure.
Fundus Photography | The procedure may be performed at all study visits (7 days and 1 month after meeting the inactivation criteria for endophthalmitis).
  Fundus imaging will be performed using the Clarus 700 Zeiss, Serial #CL700-73467, Software version 1.1.2.59261, Digital Camera Magnification 133°. Images of the posterior pole and retinal periphery will be captured, providing a comprehensive view of retinal integrity, the optic nerve, and its vasculature.

CONTACTS AND LOCATIONS:
Overall Officials: Raul Velez Montoya, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Hospital Asociación Para Evitar la Ceguera en México I.A.P., Mexico City, Mexico

DOCUMENTS (2):
  • Study Protocol (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT07175311/Prot_000.pdf
  • Informed Consent Form (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT07175311/ICF_001.pdf